CLINICAL TRIAL: NCT06361992
Title: Efficacy and Safety of Blue Cap for the Treatment of Atopic Dermatitis in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC_SERBIA_2022
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis and Related Conditions; Atopic Dermatitis Eczema; Atopic Dermatitis (AD)
Keywords: Piroctone Olamine; paediatrics; Dermatology; Atopic Dermatitis; Skin
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blue cap Foam (Experimental): Application regimen: Blue Cap foam 100 ml, Activated Piroctone Olamine (Foam, label 100 ml), Catalysis S.L. Madrid must be applied twice a day on all affected areas. The application is to be continued for 30 days, after which the patients stop using the foam until the final assessment at day 45.
  Interventions: Other: Blue Cap Foam

INTERVENTIONS:
Other: Blue Cap Foam — Application regimen: Blue Cap foam 100 ml, Activated Piroctone Olamine (Foam, label 100 ml), Catalysis S.L. Madrid must be applied twice a day on all affected areas. The application is to be continued for 30 days, after which the patients stop using the foam until the final assessment at day 45.

SUMMARY:
To verify the efficacy and tolerability of Activated Piroctone Olamine (Blue Cap Foam, label volume 100 ml) by CATALYSIS, S. L. Madrid, applied in the management of all types of dermatitis (atopic, seborrheic, eczema) in patients with significant manifestations of the disease in varying areas of the body of varying extent and to assess differences in individual tolerability and the final effect in a group of selected patients aged 3 to 18 years.

DETAILED DESCRIPTION:
The first reports on the possibility of using Activated Piroctone Olamine as an effective treatment for patients with papulosquamous dermatoses, eczema and seborrhoeic dermatitis date back to the 1970s. The observations are presented in scientific papers by dermatologists, pharmacologists and laboratory workers who have verified the original thesis in practice by the practical use of different types of products. Activated Piroctone Olamine as an active ingredient is now used by a number of companies in their product range, either as the only active ingredient or, for example, in combination with other active ingredients such as liquid carbonis detergens. The Spanish company CATALYSIS S.L Madrid has also started to produce preparations containing Activated Piroctone Olamine intended for targeted use in dermatological practice. The products have been named Blue Cap® and the original shampoo has been gradually supplemented by spray, cream and foam formulations. The company has an eminent interest in the serious evaluation of the products and has therefore ordered a number of large clinical multicentre studies carried out in different geographical zones - ranging from the Tropical, through the Temperate to the Siberian regions.

The active ingredient Activated Piroctone Olamine alone or in combination with other active ingredients makes for products with excellent properties. Activated Piroctone Olamine itself has a proven antiseptic, antimicrobial, antifungal and keratolytic effect.

The effect is selective, only acting on the morbidly altered cells. The concentrations of Activated Piroctone Olamine used in BLUE-CAP formulations are absolutely safe. The products can also be used on the surface of larger body areas and in virtually all age groups.

Activated Piroctone Olamine has a number of positive effects on pathological processes in the skin - high antimicrobial and antifungal effect, selective cytostatic effect on skin cells (at the stage of hyperproliferation, but does not affect healthy cells), it regulates the amount and number of cellular enzymes and determines the anti-inflammatory effect (if it is employed in a targeted manner in form of topically applied preparations.

To evaluate the efficacy and safety of the use of Piroctone Olamine in paediatric patients, the following clinical trial was conducted. A commercial formulation of Piroctone Olamine, Blue Cap, in foam format was used on patients aged 3 to 18 years and evaluated for safety and efficacy in the control of symptoms associated with dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Dermatitis affecting different areas of the body in varying extent.
* Outpatient status
* Age of 3 to 18 years, male, female
* Voluntary participation in the trial
* Signed informed patient consent form (Parents, legal tutor, or individual)
* One-time participation in the trial

Exclusion Criteria:

* Specific exclusion criteria

  * Usage of other systemic preparation which might influence the final assessment (natural preparations, physical therapy)
  * Known allergy to the tested preparation
  * Disease focus infection manifestations (superinfection requiring therapy)
  * Immunosuppressive therapy
  * Cancer
  * Malignancies
* General exclusion criteria:

  * Alcohol and drug abuse.
  * Participation in another clinical trial within the past 30 days.
  * Simultaneous participation in any other clinical trial.
  * Other reasons excluding the patient from the trial.
  * Restricted ability of the patient to follow therapy instructions.
  * Other physical or mental disorders disturbing the trial plan.
  * Possible consent withdrawal, presumed patient unreliability.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Grade of Patient Tolerability to the investigation product | 45 days
  Assessment of tolerance to the application of the test product in paediatric patients. This was done by following and monitoring patients in contact with the Blue Cap product at the topical level by reporting adverse effects during and after use of the product. The assessment of the tolerance of each patient is made throughout the follow-up of the patient (45 days or in case of exclusion of the patient) made by both the investigator and the patient: 1-4 (1- excellent, 2 - very good, 3 - good, 4 - intolerance).
Clinical Improvement of Patients with Dermatitis | 45 days
  Assessment of the clinical improvement of paediatric patients with dermatitis over the course of the visits using a questionnaire. The global questionnaire assesses the disappearance of clinical manifestations and improvement in skin quality with the following scale: None, Slight, Moderate, Great. The evaluation of each patient is carried out at time 0, 15 days, 30 days, 45 days or on exclusion of the patient.
Clinical assessment of symptoms and sings associated with Dermatitis | 45 days
  Evaluation of the clinical improvement of symptoms and signs associated with dermatitis in paediatric patients by means of a questionnaire on the presence or absence (Yes/No) of the following symptoms: Erythema, Scaling, Infiltration, Excoriations, Lichenification, Xerosis, Pruritus. The evaluation of each patient is carried out at time 0, 15 days, 30 days, 45 days or on exclusion of the patient.

SECONDARY OUTCOMES:
Evaluation of the therapeutic effect of Blue Cap in paediatric patients with dermatitis. | 45 days
  Evaluation of the effect of the therapy performed by the investigator according to the percentage of healing of the dermatitis affected area after the use of Blue Cap compared to baseline time: Scale of grade l-4.
  1. Excellent, 80 - 100% improvement in skin quality, excellent aesthetic effect.
  2. Satisfactory, up to 60% improvement in skin quality, satisfactory aesthetic and cosmetic effect.
  3. Insignificant improvement, 30% improvement in skin quality, dissatisfactory aesthetic and cosmetic effect
  4. Unsatisfactory condition, finding in original extent.
Evaluation of the therapeutic effect of Blue Cap on healing of the skin at the patients | 45 days
  Subjective evaluation of the effect of the therapy on skin healing by the investigator visually based on the healing of the dermatitis affected area after use of Blue Cap compared to baseline time: Scale of grade l - 4.
  1. Excellent aesthetic and cosmetic effect, no undesired effects
  2. Satisfactory aesthetic effect
  3. Insignificant improvement, unsatisfactory effect
  4. Unsatisfactory effect

CONTACTS AND LOCATIONS:
Locations (3):
- Serbia (3):
  - University of Niš Faculty of Medicine, Department of Dermatology and Venereology, University Clinical Center of Niš, Niš, Nišava
  - City Institute for Skin and Venereal Diseases Belgrade, Belgrade
  - University of Belgrade Faculty of Medicine, University Clinical Center of Serbia, Belgrade

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Background] Leung DY. New insights into atopic dermatitis: role of skin barrier and immune dysregulation. Allergol Int. 2013 Jun;62(2):151-61. doi: 10.2332/allergolint.13-RAI-0564. PMID 23712284
- [Background] Chovatiya R, Paller AS. JAK inhibitors in the treatment of atopic dermatitis. J Allergy Clin Immunol. 2021 Oct;148(4):927-940. doi: 10.1016/j.jaci.2021.08.009. Epub 2021 Aug 24. PMID 34437922
- [Background] Hamilton JD, Suarez-Farinas M, Dhingra N, Cardinale I, Li X, Kostic A, Ming JE, Radin AR, Krueger JG, Graham N, Yancopoulos GD, Pirozzi G, Guttman-Yassky E. Dupilumab improves the molecular signature in skin of patients with moderate-to-severe atopic dermatitis. J Allergy Clin Immunol. 2014 Dec;134(6):1293-1300. doi: 10.1016/j.jaci.2014.10.013. PMID 25482871
- [Background] Nakashima C, Yanagihara S, Otsuka A. Innovation in the treatment of atopic dermatitis: Emerging topical and oral Janus kinase inhibitors. Allergol Int. 2022 Jan;71(1):40-46. doi: 10.1016/j.alit.2021.10.004. Epub 2021 Nov 21. PMID 34815171
- [Background] Puviani M, Campione E, Offidani AM, De Grandi R, Bianchi L, Bobyr I, Giannoni M, Campanati A, Bottagisio M, Bidossi A, De Vecchi E, Eisendle K, Milani M. Effects of a cream containing 5% hyaluronic acid mixed with a bacterial-wall-derived glycoprotein, glycyrretinic acid, piroctone olamine and climbazole on signs, symptoms and skin bacterial microbiota in subjects with seborrheic dermatitis of the face. Clin Cosmet Investig Dermatol. 2019 May 2;12:285-293. doi: 10.2147/CCID.S205904. eCollection 2019. PMID 31190937
- [Background] Piquero-Casals J, Hexsel D, Mir-Bonafe JF, Rozas-Munoz E. Topical Non-Pharmacological Treatment for Facial Seborrheic Dermatitis. Dermatol Ther (Heidelb). 2019 Sep;9(3):469-477. doi: 10.1007/s13555-019-00319-0. Epub 2019 Aug 8. PMID 31396944
- [Background] Pierard-Franchimont C, Goffin V, Henry F, Uhoda I, Braham C, Pierard GE. Nudging hair shedding by antidandruff shampoos. A comparison of 1% ketoconazole, 1% piroctone olamine and 1% zinc pyrithione formulations. Int J Cosmet Sci. 2002 Oct;24(5):249-56. doi: 10.1046/j.1467-2494.2002.00145.x. PMID 18498517
- [Background] Fabbrocini G, Panariello L, DE Padova MP, Lorenzi S, Caro G, Marasca C, Russo G. Efficacy and tolerability of a spray product containing hydroxypropyl chitosan, climbazole and piroctone olamine, applied twice weekly for the treatment of the pitiriasis versicolor. G Ital Dermatol Venereol. 2017 Dec;152(6):565-568. doi: 10.23736/S0392-0488.16.05299-8. Epub 2016 Jul 5. PMID 27377141
- See also: Results of the pilot study conducted with Blue Cap Foam in paediatric patients previously in Slovakia. — https://www.kosmetischemedizin-online.de/case-study/abschlussbericht-ueber-die-pilotstudie-zur-ueberpruefung-der-wirkung-von-activated-piroctone-olamine-etikett-100ml-bei-der-behandlung-von-psoriasis-und-seborrhoischer-dermatitis-bei-patienten-im-alt/
- See also: Results of the pilot study conducted with Blue Cap Foam in paediatric patients previously in St. Petersburg. — https://pediatria.orscience.ru/2658-6630/article/view/111070